CLINICAL TRIAL: NCT06648850
Title: Clinical Study of DA-001 as a Treatment for Hair Shedding Reduction and Hair Re-Growth
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Applied Biology, Inc. (Industry)
Collaborators: Follea International Limited (Industry); Daniel Alain, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DA-001-TE
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Telogen Effluvium; Female Pattern Hair Loss; Female Pattern Hair Loss, Androgenic Alopecia
Keywords: Hair Shedding; hair growth
MeSH Terms: conditions — Alopecia | interventions — Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- DA-001 Topical (Experimental): Phenylephrine 2.5% Topical + TAAR agonist
  Interventions: Drug: DA-001
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- Phenylephrine Topical (Experimental): Phenylephrine 2.5% Topical
  Interventions: Drug: Phenylephrine
- DA-001 Topical + DA-005 Oral (HIF-1α supplement) (Experimental): DA-001 Topical (Phenylephrine 2.5% Topical + TAAR agonist tyramine) + DA-005 Oral (HIF-1α supplement)
  Interventions: Other: DA-001 Topical + DA-005 Oral (HIF-1α supplement)
- DA-010 - Oral Phenylephrine 20 mg + DA-005 Oral (HIF-1α supplement) (Experimental): Oral Phenylephrine 20 mg + DA-005 Oral (HIF-1α supplement)
  Interventions: Drug: DA-010 - Oral Phenylephrine 20 mg + DA-005 Oral (HIF-1α supplement)

INTERVENTIONS:
Drug: DA-001 — Phenylephrine 2.5% Topical + TAAR Agonist (GRAS) Topical Solution
  Arms: DA-001 Topical
Other: Placebo — Placebo Topical Solution
  Arms: Placebo
Drug: Phenylephrine — Phenylephrine 2.5% Topical
  Arms: Phenylephrine Topical
Other: DA-001 Topical + DA-005 Oral (HIF-1α supplement) — DA-001 Topical (Phenylephrine 2.5% Topical + TAAR agonist tyramine) + DA-005 Oral (HIF-1α supplement)
  Arms: DA-001 Topical + DA-005 Oral (HIF-1α supplement)
Drug: DA-010 - Oral Phenylephrine 20 mg + DA-005 Oral (HIF-1α supplement) — Oral Phenylephrine 20 mg + DA-005 Oral (HIF-1α supplement)
  Arms: DA-010 - Oral Phenylephrine 20 mg + DA-005 Oral (HIF-1α supplement)

SUMMARY:
The primary objective of the study is to assess the safety and efficacy of DA-001 as a treatment for Hair Shedding Reduction and Hair Re-Growth

DETAILED DESCRIPTION:
DA-001 is a topical alpha 1 agonist combined with a TAAR receptor agonist. DA-001 was studied in a population of women that suffer from excessive hair shedding. DA-001 demonstrated significant reduction in hair shedding.

This study aims to assess the safety and efficacy of DA-001 as a treatment for Hair Shedding Reduction and Hair Re-Growth.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Diagnosed with telogen effluvium
* Willing and able to apply the treatment as directed, comply with study
* Otherwise healthy
* Able to give informed consent

Exclusion Criteria:

* A medical history that may interfere with study objectives
* Women who are pregnant, lactating, or planning to become pregnant during the study period
* Subjects who have experienced a clinically important medical event within 90 days of the visit (e.g., stroke, myocardial infarction, etc)
* Subjects who have known allergies to any excipient in DA-001
* Subjects who are currently participating in another clinical study or have completed another clinical study with an investigational drug or device in the treatment area within 30 days prior to study treatment initiation
* Subjects who have used any topical prescription medications in the treatment area within 30 days prior to study treatment initiation
* Subjects who have had a dermatological procedure such as surgery in the treatment area within 30 days prior to study treatment initiation
* Subject is unable to provide consent or make the allotted clinical visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2027-02-19 (Estimated); Study Completion 2027-03-26 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Hair Shedding | Minutes [0,5]
  Number of hairs shedding during brushing at target area

SECONDARY OUTCOMES:
Mean Change in Hair Shedding | Week [0, 4, 12, 24]
  Number of hairs shedding during brushing at target area
Mean Change in Target Area Hair Count (TAHC) | Week [0, 4, 12, 24]
  Number of hairs in a 1-cm² target scalp area

CONTACTS AND LOCATIONS:
Overall Officials: Andy Goren, MD, Study Director — University of Rome G. Marconi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Daniel Alain, Inc. - Updated Study Information — http://www.danielalain.com